CLINICAL TRIAL: NCT06172400
Title: Wide Awake Open Carpal Tunnel Release With or Without a Tourniquet: a Randomized Single-blinded Controlled Trial
Brief Title: Wide Awake Open Carpal Tunnel Release With or Without a Tourniquet
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Region Skane (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2020-04670
Record Dates: First submitted 2023-12-07; First posted 2023-12-15 (Actual); Last update posted 2023-12-26 (Actual); Status verified 2023-12

CONDITIONS: Carpal Tunnel Syndrome
MeSH Terms: conditions — Carpal Tunnel Syndrome | interventions — Mepivacaine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Touniquet (Active Comparator): Local injection of Mepivacaine (10 mg/ml) approximately 10 ml in the incisional area at least 10 minutes before surgery start. Use of a forearm tourniquet at the pressure of 250 mmHg.
  Interventions: Drug: Mepivacaine, Combinations
- Adrenaline (Experimental): Local injection of Mepivacaine (10 mg/ml) and adrenaline (5 mcg/ml) approximately 10 ml in the incisional area at least 10 minutes before surgery start. Forearm tourniquet applied but not inflated.
  Interventions: Drug: Mepivacaine, Combinations

INTERVENTIONS:
Drug: Mepivacaine, Combinations — Using local anesthesia with adrenaline for intraoperative vasoconstriction instead of a tourniquet.

SUMMARY:
The goal of this clinical trial is to compare open carpal tunnel release using local anesthesia with or without a tourniquet. The main questions it aims to answer are:

1. Do the tourniquet cause more procedural pain?
2. Does the use of tourniquet affect the outcome after the procedure? Participants will be randomized to either local anesthesia with a tourniquet or local anesthesia with adrenaline, and undrgo standard open carpal tunnel release.

ELIGIBILITY:
Inclusion Criteria:

* Primary idiopathic CTS
* Age 18 or older
* Symptoms of classic or probable carpal tunnel syndrome according to Katz hand diagram
* No previous wide awake hand surgical procedures under local anesthesia
* No planned concomitant procedures

Exclusion Criteria:

* Recurrent carpal tunnel syndrome
* Vibration induced neuropathy
* Polyneuropathy
* Cognitive impairment
* Anxiety disorder
* Swedish language insufficiency
* Active substance abuse
* Allergy to local anesthesia or adrenaline
* Patient refusal to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-01-09 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Procedural pain | Day 1
  Visual analog scale 0 (no pain)-100 (worst possible pain)

SECONDARY OUTCOMES:
Injection pain | Day 1
  Visual analog scale 0 (no pain)-100 (worst possible pain)
Procedure satisfaction | Day 1
  Visual analog scale 0 (best)-100 (worst)
Surgery time | Day 1
  Incision to wound closure (minutes)
Use of diathermy/need to inflate or deflate tourniquet | Day 1
Adverse events | 2 weeks
11-item disabilities of arm, shoulder and hand questionnaire (QuickDASH) | 3 months, 1 year
  0 (best)-100 (worse)
Atroshi-Lyrén scale | 3 months, 1 year
  1 (no symptoms)- 5 (worst symptoms)
Palmar pain scale | 3 months, 1 year
  0 (no palmar pain or activity limitation)-100 (worst)

IPD SHARING:
Plan to Share IPD: No